CLINICAL TRIAL: NCT05707247
Title: Evaluation of the Feasibility of an Expert Decision Support System for Patients Regarding the Optimization of the Management of Drugs With Conditional Administration in the Surgical Department: Pilot Study
Brief Title: Study of a Prototype Software to Help Surgical Patients Manage Their Pain Medication
Acronym: MORPHEE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 8706
Record Dates: First submitted 2023-01-12; First posted 2023-01-31 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Post-operative Situation
Keywords: prototype software; patient interface; experimental medical device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prototype software (Experimental)
  Interventions: Device: software

INTERVENTIONS:
Device: software — The experimental medical device is a prototype software. It is a patient interface.
  The device comes in the form of a smartphone with a touch screen

SUMMARY:
The experimental medical device is a prototype software. The device comes in the form of a smartphone with a touch interface. The smartphone used to support the software is a commercial smartphone marked CE. The study aims at assessing the feasibility of the use of this expert, patient- decision support systems.

The study hypothesis is that the clinical use of the experimental device is feasible.

ELIGIBILITY:
Inclusion criteria:

* Male or Female 18 years or older (no upper age limit)
* Operated within a surgical department of of the Hautepierre University Hospitals of Strasbourg
* Patient understanding and reading French
* Subject neurosensorially able of interacting with a tactile electronical interface
* Subject able to understand research objectives, risks and provide dated and signed informed consent
* Subject covered by a health insurance scheme

Exclusion criteria:

* Patient with neuropsychiatric or sensory disorders that may interfere with their use of the visual interface
* Unable to provide informed information (subject in emergency, difficulty understanding the subject, etc.)
* Pregnant or lactating woman (on declaration)
* Patient under safeguard of justice, under guardianship, under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of the INSAMED computer tool | Day 2 post operative
  agreement between INSAMED computer tool and the recommendations established by caregivers. The data from INSAMED computer tool will be collected by extracting the history of the digital interface (commercial smartphone) hosting the expert system.

SECONDARY OUTCOMES:
Evaluate the time delay, in usual care setting, of rescue drug administrations after surgery, to confirm the interest of developing expert systems to improve the existing one. | 60 minutes after software activation
  Delay, in minutes, between soliciting a ward nurse as usual practice (e.g., doorbell) and the administration of the therapeutic response.
  This time will be collected by the Research IDE during patient interview. 60 minutes after software activation. The patient will simultaneously request the standard care IDE (doorbell) and the INSAMED tool.
Assess patient satisfaction with usual care | 60 minutes after software activation.
  Patient satisfaction with the routine care therapeutic response measured by an analog visual scale between 0 and 100, measured 60 minutes after software activation.
Assess patient satisfaction with the ease of use of the experimental device | 60 minutes after software activation.
  Patient satisfaction with the ease of use of the INSAMED device measured by an analog visual scale between 0 and 100, measured 60 minutes after software activation
assess the security of the device | Day 2 post operative
  Safety analysis of INSAMED software through evaluation of serious adverse events based on a expert panel reviewing.

CONTACTS AND LOCATIONS:
Overall Officials: Eric NOLL, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Background] Noll E, Noll-Burgin M, Bonnomet F, Reiter-Schatz A, Gourieux B, Bennett-Guerrero E, Goetsch T, Meyer N, Pottecher J. Knowledge-based, computerized, patient clinical decision support system for perioperative pain, nausea and constipation management: a clinical feasibility study. J Clin Monit Comput. 2024 Aug;38(4):907-913. doi: 10.1007/s10877-024-01148-z. Epub 2024 Apr 12. PMID 38609723